CLINICAL TRIAL: NCT03695705
Title: Randomized Control Trial of Rifaximin and Norfloxacin in Primary and Secondary Prophylaxis of Spontaneous Bacterial Peritonitis(SBP) in Cirrhotic Patients
Brief Title: Rifaximin and Norfloxacin for Prevention of SBP in Adults With Decompensated Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Radha K Dhiman, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PGIMER
Record Dates: First submitted 2018-09-27; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Cirrhosis, Liver
Keywords: Norfloxacin,Rifaximin,Prophylaxis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Rifaximin; Norfloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary prophylaxis arm (Other): 28 Patients with decompensated cirrhosis without past history of SBP were randomised to receive Rifaximin at dose 550 mg twice daily.29 Patients with decompensated cirrhosis without past history of SBP were randomized to receive Norfloxacin at dose 400 mg once daily
  Interventions: Drug: Rifaximin 550 mg twice a day and Norfloxacin 400 mg once a day
- Secondary prophylaxis arm (Other): 26 Patients with decompensated cirrhosis with past history of SBP were randomized to receive Rifaximin at dose 550 mg twice daily.33 Patients with decompensated cirrhosis with past history of SBP were randomized to receive Norfloxacin at dose 400 mg once daily
  Interventions: Drug: Rifaximin 550 mg twice a day and Norfloxacin 400 mg once a day

INTERVENTIONS:
Drug: Rifaximin 550 mg twice a day and Norfloxacin 400 mg once a day — Patients on Rifaximin prophylaxis will be given 550 mg twice daily and on Norfloxacin prophylaxis will receive Norfloxacin 400 mg once daily for 6 months

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is a frequent and severe complication of cirrhotic patients with ascites.Early diagnosis and prompt treatment with effective antibiotics significantly improves the prognosis of this complication. The recommended treatment is a third generation cephalosporin given intravenously for five days.Following recovery patients should receive secondary prophylaxis with a quinolone such as oral norfloxacin 400 mg/day.Also all patients should be assessed for liver transplantation.

Most commonly used antibiotic for both primary and secondary prophylaxis is norfloxacin 400 mg once daily.Other antibiotics like cotrimoxazole,ceftriaxone,ciprofloxacin and rifaximin have also been evaluated in various studies.Use of antibiotic prophylaxis has been evaluated to decrease recurrence of SBP in treated groups than in control groups.

Rifaximin is an oral antimicrobial agent with broad-spectrum activity that is gut-selective and nonsystemic. Rifaximin appears to have a low level of selection for resistant bacterial mutants. Intestinal decontamination is known to increase peripheral blood counts by suppressing endotoxemia and inhibiting the effects of cytokines and nitric oxide on blood counts.

With this mechanisms rifaximin has been already proven to decrease recurrence of hepatic encephalopathy.The most important mechanism for development of SBP is bacterial translocation (BT).Translocation of enteric flora occurs via defective mucosal barrier.BT is considered the key step in pathogenesis of SBP and cirrhotic patients.It is also the critical factor that is responsible for host immune response and secreation of inflammatory mediators that is responsible for hemodynamic changes in cirrhotics.Three most important mechanism of bacterial translocation include bacterial overgrowth,physical disruption of gut mucosal barrier and impaired host defence.

Rifaximin by mechanism of gut decontamination may reduce translocation of intestinal bacteria into mesenteric lymph nodes then into ascitic fluid.Thus it may prove useful in preventing recurrence of SBP.There was no study till date that has compared efficacy of Norfloxacin and rifaximin to prevent development of SBP.This pilot study was done to compare the efficacy of rifaximin with norfloxacin in both primary and secondary prophylaxis of SBP in a prospective randomized open-label and non-inferiority trial

DETAILED DESCRIPTION:
Ascites is the most common complication of cirrhosis, and 60% of patients with compensated cirrhosis develop ascites within 10 years during the course of their disease . Ascites occurs only when portal hypertension has developed and is related to inability to excrete an adequate amount of sodium into urine, leading to a positive sodium balance.Evidence suggests that renal sodium retention in patients with cirrhosis is secondary to arterial splanchnic vasodilation. This causes a decrease in effective arterial blood volume with activation of arterial and cardiopulmonary volume receptors, and homeostatic activation of vasoconstrictor and sodium-retaining systems (i.e., the sympathetic nervous system and the (renin-angiotensin-aldosterone system). Renal sodium retention leads to expansion of the extracellular fluid volume and formation of ascites and edema . The development of ascites is associated with a poor prognosis and impaired quality of life in patients with cirrhosis . Thus, patients with ascites should generally be considered for referral for liver transplantation. There is a clear rationale for the management of ascites in patients with cirrhosis, as a successful treatment may improve the outcome and symptoms.

Spontaneous bacterial peritonitis (SBP) is a frequent and severe complication of cirrhotic patients with ascites.Early diagnosis and prompt treatment with effective antibiotics significantly improves the prognosis of this complication. The recommended treatment is a third generation cephalosporin given intravenously for five days. The most commonly used is cefotaxime, up to 4 g/day in 2-4 divided doses because of its proven efficacy and safety3. Repeat diagnostic paracentesis to document response by a greater than 25% decrease in ascitic fluid neutrophil count at 48 hours after commencement of antibiotic is recommended. With this regimen, recovery from SBP is higher than 80-90% and 30-day survival is at least 80%.Following recovery patients should receive secondary prophylaxis with a quinolone such as oral norfloxacin 400 mg/day.Also all patients should be assessed for liver transplantation

.Most commonly used antibiotic for both primary and secondary prophylaxis is norfloxacin 400 mg once daily.Other antibiotics like cotrimoxazole,ceftriaxone,ciprofloxacin and rifaximin have also been evaluated in various studies.Use of antibiotic prophylaxis has been evaluated to decrease recurrence of SBP in treated groups than in control groups.

Rifaximin is an oral antimicrobial agent with broad-spectrum activity that is gut-selective and nonsystemic. Rifaximin appears to have a low level of selection for resistant bacterial mutants and may not confer the same risks as those associated with systemic antibiotics. A study in patients with alcohol-related decompensated cirrhosis reported that rifaximin treatment reduced endotoxin levels and resulted in significantly decreased hepatic venous pressure gradient values, which decreased the occurrence of complications in advanced liver disease.13Intestinal decontamination with rifaximin has been shown to increase platelet count significantly in thrombocytopenic patients with cirrhosis.This benefit is thought to be achieved through a concomitant reduction of endotoxemia.Improvements in platelet counts in patients with thrombocytopenia could decrease bleeding risks and complications of medical procedures, and help stabilize underlying liver disease. Intestinal decontamination is also known to increase peripheral blood counts by suppressing endotoxemia and inhibiting the effects of cytokines and nitric oxide on blood counts.

With this mechanisms rifaximin has been already proven to decrease recurrence of hepatic encephalopathy.The most important mechanism for development of SBP is bacterial translocation (BT) which refers to entry of bacteria or their products into regional lymph nodes,systemic circulation and extraintestinal organs.Translocation of enteric flora occurs via defective mucosal barrier.BT is considered the key step in pathogenesis of SBP and cirrhotic patients.It is also the critical factor that is responsible for host immune response and secreation of inflammatory mediators that is responsible for hemodynamic changes in cirrhotics.Three most important mechanism of bacterial translocation include bacterial overgrowth,physical disruption of gut mucosal barrier and impaired host defence.

Rifaximin by mechanism of gut decontamination may reduce translocation of intestinal bacteria into mesenteric lymph nodes then into ascitic fluid.Thus it may prove useful in preventing recurrence of SBP.There is no study till date that has compared efficacy of Norfloxacin and rifaximin to prevent development of SBP.This pilot study was done to compare the efficacy of rifaximin with norfloxacin in both primary and secondary prophylaxis of SBP in a prospective randomized open-label and non-inferiority trial

ELIGIBILITY:
Inclusion Criteria:

1. Low Ascitic fluid protein level <1gm/dl
2. Advanced liver disease as evidenced by CTP≥9
3. Serum billirubin≥3 mg/dl
4. Impaired renal function defined by serum creatinine≥1.2 mg/dl
5. Blood urea nitrogen 25mg/dl
6. Serum sodium level≤ 1.2 meq/l

Exclusion Criteria:

1. Inability to obtain informed consent from patient or relatives.
2. Acute on chronic liver failure
3. Severe cardiopulmonary disease
4. Pregnancy
5. Age <18yrs
6. Post liver transplant patients
7. HIV infection
8. Recent abdominal surgery(with in last 6 months)
9. Portal vein thrombosis
10. Splenectomy
11. Patient on immunosuppressive drugs except for alcoholic steatohepatitis
12. Patients on psychoactive drugs, such as antidepressants or sedatives
13. Hypersensitivity to norfloxacin and rifaximin
14. Malignancies including Hepatocellular carcinoma
15. Prior history of hepatic encephalopathy on Rifaximin -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence SBP in patients on Rifaximin prophylaxis compared to Norfloxacin | 6 months
  Incidence of development of SBP in patients with(Secondary prophylaxis) or without(Primary prophylaxis) in patients on Rifaximin compared to norfloxacin

SECONDARY OUTCOMES:
Incidence of hepatic encephalopathy | 6 months
  Incidence of development of hepatic encephalopathy in patients on Rifaximin prophylaxis compared to Norfloxacin prophylaxis
Incidence of overall mortality | 6 months
  Incidence of mortality in patients on Rifaximin prophylaxis compared to Norfloxacin prophylaxis
Incidence of development of sepsis | 6 months
  Incidence of development of sepsis in patients on Rifaximin prophylaxis compared to Norfloxacin prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: RADHA K DHIMAN, DM,FRCP, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Praharaj DL, Premkumar M, Roy A, Verma N, Taneja S, Duseja A, Dhiman RK. Rifaximin Vs. Norfloxacin for Spontaneous Bacterial Peritonitis Prophylaxis: A Randomized Controlled Trial. J Clin Exp Hepatol. 2022 Mar-Apr;12(2):336-342. doi: 10.1016/j.jceh.2021.08.010. Epub 2021 Aug 18. PMID 35535057